CLINICAL TRIAL: NCT02800538
Title: The Effects of Intragastric Administration of Nutrients on Executive Control in Healthy Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S56123
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2016-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lauric acid (Experimental): the nutrient that can be widely found in daily food.
  Interventions: Dietary Supplement: intragastric infusion of nutrient
- Palmitic acid (Experimental): the nutrient that can be widely found in daily food.
  Interventions: Dietary Supplement: intragastric infusion of nutrient
- Capric acid (Experimental): the nutrient that can be widely found in daily food.
  Interventions: Dietary Supplement: intragastric infusion of nutrient
- Saline (Placebo Comparator): physiological salt water
  Interventions: Dietary Supplement: intragastric infusion of nutrient

INTERVENTIONS:
Dietary Supplement: intragastric infusion of nutrient — Intragastric infusion of nutrient that can be widely found in daily food or placebo.

SUMMARY:
The previous research by one of our members in the research team (H. Miller) suggests a possible influence of oral nutrients intake of certain fat or carbohydrates (glucose, fructose) on executive control. On the other hand, another previous study from our group (L. Van Oudenhove) suggests a subliminal influence of intragastric administration of fatty acids on subjective and neural responses to negative emotion induction. The purpose of this study therefore is to examine the effect of intragastric administration of certain fatty acids and carbohydrates on executive control in healthy volunteers.

Therefore one group of healthy volunteers are invited to the study. The participants will be randomly administered one of the three fatty acid emulsions or placebo via a nasogastric tube in each of the visits. After the exposure period, participants will use a computer to perform there different tasks to measure executive control. During each study visit, regular measurements of emotion, physical sensations, as well as blood glucose will be assessed. Furthermore, an electrocardiogram will be continuously recorded for the calculation of vagal function.

ELIGIBILITY:
Inclusion Criteria:

* N = 26 These numbers are based on a power calculation for a repeated measures ANOVA with one within-subject factor using Gpower software version 3.1.7 (http://www.psycho.uni-duesseldorf.de/abteilungen/aap/gpower3), indicating that these sample sizes are needed to achieve 90% power to detect a medium-sized effect (f = 0.25).
* Men & women
* Age: >17 years
* 20 ≤ BMI ≤ 25
* Of good mental and physical health

Exclusion Criteria:

Participants with one or more of self-reported points below will be excluded:

1. History of, or current presence of:

   * Psychiatric disorders (e.g., anxiety disorders, somatization disorder, eating disorders, depression, substance-related disorders alcohol abuse or dependence etc.)
   * Abnormal eating behavior (including restraint and emotional eating)
   * Abdominal/thoracic surgery
   * Neurological, endocrine or digestive related disorders
   * Head trauma with loss of consciousness
   * Other serious medical conditions
   * Use of any drugs, including cannabis, during the past 6 months
2. Current presence of:

   * Pregnancy
   * Medication use that affects the function of the gastrointestinal tract and/or affects the nervous system, psychotropics or painkillers
   * A recent accident or surgery that has not fully recovered
3. Other

   * Smoking
   * Women not taking hormonal contraception

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
trial making task | 60 min after intervention
  Participants will be required to connect a set of 25 numbered dots in numerical order as fast as possible while still maintaining accuracy.
digital span task | 60 min after intervention
  Participants will be presented with a series of single-digit numbers and required to remember them. After the series has been presented the participants will need to indicate the numbers presented.
memory task | 60 min after intervention
  A list of 15 words that are matched for frequency, concreteness, and imagery will be presented to the participant via a computer monitor at the rate of one every 2 sec. Afterwards they will be given 60 sec to write down as many words as they are able to recall from the list. Accuracy and errors will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Belgium